CLINICAL TRIAL: NCT00271947
Title: Crohn's Disease Non-myeloablative Autologous Hematopoietic Stem Cell Transplantation (CDNST) Versus Standard Therapy
Brief Title: Crohn's Disease Stem Cell Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The PI, who was sponsor got retired
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Richard Burt, MD, MD, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD Randomized
Record Dates: First submitted 2006-01-02; First posted 2006-01-04 (Estimated); Results first posted 2014-03-27 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-02

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologous Stem Cell Transplantation (Experimental): Autologous Stem Cell Transplantation will be performed after the conditioning regimen
  Interventions: Biological: Autologous Stem Cell Transplantation

INTERVENTIONS:
Biological: Autologous Stem Cell Transplantation — Autologous Stem Cell Transplantation will be performed after conditioning regimen

SUMMARY:
Crohn's disease (CD) is a chronic illness, immunologically mediated, probably induced by the exposure of the intestine to an antigen or antigens similar to the intestine, to which immunologic tolerance is lost or a dysregulated immunity ensues. The disease has a variable course, from a mild, intermittently active illness requiring only symptomatic therapy to a fulminant illness requiring potentially dangerous immunosuppressive therapy, surgery or both. The molecular defect causing CD has not been characterized, but probably involves aberrant T cell function. Although CD often responds to immunosuppressive medication including corticosteroids, azathioprine and 6-mercaptopurine, to anti inflammatory drugs such as 5 aminosalicylate (5 ASA), or to some antimicrobial agents, including metronidazole, no therapy has been curative. In patients with severe CD, who have been unresponsive to corticosteroids, azathioprine, 5 ASA, metronidazole, and infliximab, we propose to compare the efficacy of Crohn's disease non-myeloablative autologous hematopoietic stem cell transplantation (CDNST) to standard therapy. Subsequent disease activity will be followed by (1) Crohn's disease activity index (CDAI), (2) a more global severity index, the Crohn's Severity Index, (3) type and amount of therapy for CD, and (4) clinical, hematologic and biochemical studies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older and less than age 55 years at time of pretransplant evaluation.
* An established clinical diagnosis of severe CD that has failed therapy with prednisone, azathioprine, 5 ASA products and metronidazole, and has failed an anti-TNF alpha inhibitor. Failure is defined as a CDAI (appendix A) 225-400.
* Pre-study peripheral blood counts must include a platelet count greater than 100,000/ul and an absolute neutrophil count greater than 1500/ul.
* In those randomized to receive the transplant, a stem cell harvest greater than 2.0 x 106 CD34 cells/kg is required.
* Ability to give informed consent.

Exclusion Criteria:

* HIV positive.
* History of coronary artery disease, or congestive heart failure.
* Uncontrolled diabetes mellitus, or any other illness that in the opinion of the investigators would jeopardize the ability of the patient to tolerate aggressive chemotherapy.
* Prior history of malignancy except localized basal cell or squamous skin cancer. Other malignancies for which the patient is judged to be cured by local surgical therapy, such as head and neck cancer, or stage I breast cancer will be considered on an individual basis.
* Positive pregnancy test, lactation, inability or unwillingness to pursue effective means of birth control, failure to accept or comprehend irreversible sterility as a side effect of therapy.
* Psychiatric illness or mental deficiency making compliance with treatment or informed consent impossible.
* FEV 1/FVC < 50% of predicted, DLCO < 50% of predicted.
* Resting LVEF < 40%.
* Bilirubin > 2.0 mg/dl, transferase (AST) > 2x upper limit of normal.
* Serum creatinine > 2.0 mg/dl.
* Platelet count less than 100,000/ul, ANC less than 1500/ul.
* Patients presenting with intestinal perforation or toxic megacolon, or a suppurative problem that will require urgent surgery. In addition, the patient may not have any active infection. The presence of intestinal stomas does not exclude the patient from study.
* Splenomegaly (palpable spleen on physical exam).
* Inability to collect > 2.0 x 106 CD34+ cells/kg.
* Positive pregnancy test.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2005-04; Primary Completion 2012-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Craig, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Feinberg School of Medicine, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: enrolled (n=1)
Groups:
- Autologous Stem Cell Transplantation: stem cell transplantation : Autologous Hematopoietic Stem Cell Transplantation will be performed after conditioning regimen
Period: Overall Study
Arm/Group | Autologous Stem Cell Transplantation
Started | 1
Completed | 0
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Stem Cell Transplantation: stem cell transplantation : Autologous Hematopoietic Stem Cell Transplantation will be performed on all participants randomized to transplant arm.
Arm/Group | Stem Cell Transplantation
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Remission or Clinical Improvement as Assessed by Crohn's Disease Activity Index (CDAI) Scores
Description: Clinical remission defined as a CDAI less than 150 and clinical improvement defined as decline in CDI> or = 70 one year following entry. The participant was not assessed according to the criteria of the outcome measure, because the participant was lost for follow-up.
Time Frame: baseline
Arm/Group | Stem Cell Transplantation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: CDAI
Arm/Group | Stem Cell Transplantation
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Potential participants refused to be randomized. Just one participant was enrolled on study, the study is terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes